CLINICAL TRIAL: NCT03909542
Title: Postoperative Complications in Patients With Inflammatory Bowel Disease: A Retrospective Cohort Study
Brief Title: Malnutrition Associated With Complications After Ileostomy Reversal
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joel Bauer, Dr. Joel J Bauer MD, Professor of Surgery, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 16-0139
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Inflammatory Bowel Diseases; Ileostomy
Keywords: inflammatory bowel disease; ileostomy; ileostomy reversal; stoma reversal
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ileostomy Closure: Patients who have undergone an ileostomy closure procedure.

SUMMARY:
An ileostomy is a surgical opening established by bringing the end or a loop of the ileum to discharge directly outside the body. This is typically done when part or the entire colon is removed because of IBD, cancer, or familial adenomatous polyposis. Reversal of this procedure, an ileostomy closure, may be done if possible. Ileostomy closure involves reconnecting the ileum to the remaining colon, allowing normal bowel movements again. This study will look at the outcomes of these surgeries in patients who were seen and operated on by the investigators.

DETAILED DESCRIPTION:
This study focused on outcomes and complications after ileostomy closure. An ileostomy is a surgical opening established by bringing the end or a loop of the ileum to discharge directly outside the body. This is typically done when part or the entire colon is removed because of IBD, cancer, or familial adenomatous polyposis. Reversal of this procedure, an ileostomy closure, may be done if possible to reconnect the ileum to the remaining colon and allow normal bowel movements again. This study looked at the outcomes for these surgeries in patients who were seen and operated on by the investigators. Patients were identified from the files and schedules of the investigators, and Epic was used to collect the information needed to determine perioperative clinical characteristics and post-operative outcomes. This data was kept in a secure electronic database, with identifiers removed as soon as all of the data was collected for a patient.

ELIGIBILITY:
Inclusion Criteria:

* ileostomy closure procedure

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have had an ileostomy closure procedure
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Number of Complications | up to 5 years
  Number of any post operative complication

CONTACTS AND LOCATIONS:
Overall Officials: Joel J Bauer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No